CLINICAL TRIAL: NCT02676765
Title: Desensitization and Cross-Desensitization During Oral Grass or Ragweed Pollen Immunotherapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Intellectual property issues with drug manufacture.
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: HM20006291; MISP 52707 (Other Grant/Funding Number: Merck)
Record Dates: First submitted 2016-02-03; First posted 2016-02-08 (Estimated); Results first posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-02

CONDITIONS: Immunologic Desensitization
Keywords: Allergic rhinitis; Immunotherapy, Allergen; Sublingual Immunotherapy
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Allergens

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- sublingual allergen tablets (Experimental): Subjects will be administered a sublingual allergen tablet customized to their individual allergic sensitization.
  Interventions: Drug: allergen extract tablet
- Placebo (Placebo Comparator): Subjects will be administered placebo sublingual tablets
  Interventions: Drug: Placebo tablet

INTERVENTIONS:
Drug: allergen extract tablet — 1 allergen extract tablet, placed under the tongue until dissolved, taken daily; do not swallow for 1 minute after placing tablet; do not eat or drink for 5 minutes after placing tablet
  Other Names: Ragwitek; Grastek
  Arms: sublingual allergen tablets
Drug: Placebo tablet — 1 placebo tablet, placed under the tongue until dissolved, taken daily; do not swallow for 1 minute after placing tablet; do not eat or drink for 5 minutes after placing tablet
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if sublingual allergen immunotherapy tablets work by inducing a state of desensitization in mast cells and basophils.

DETAILED DESCRIPTION:
To induce clinical tolerance, a failure to respond to an allergen to which one was previously responsive, is an important objective for physicians, one that plays a significant role in the primary prevention of allergic reactions in the clinical practice of Allergy & Immunology. The tolerance resulting after standard subcutaneous immunotherapy to aeroallergen and insect venom allergens is long lasting and allergen-specific, and may involve antigen-specific T regulatory cells. In contrast, tolerance resulting from drug desensitization protocols is short-lived, and postulated to target mast cells and basophils. Research into the cellular and biochemical processes by which desensitization occurs has revealed that mast cells desensitized to one antigen in vitro, under certain conditions, lose the ability to degranulate to unrelated antigens or to direct FcεRI cross-linking. Preliminary data suggests that this cross-desensitization can happen in patients undergoing incremental desensitization, depending in part on the percentage of IgE targeted to the allergen used for desensitization. This proposal therefore aims to explore desensitization and cross-desensitization in human volunteers undergoing standard sublingual (SL) immunotherapy to grass or ragweed pollen.

Subjects will undergo SL immunotherapy with either Timothy or Short Ragweed tablets, taking one tablet per day, or will take a placebo tablet. Titration skin testing to Timothy or Short Ragweed, to one or preferably two additional allergens to which the subject is sensitive, and to codeine as a control for mast cell activation capability through a non-IgE-dependent pathway will be performed to determine the PC3 value (see below). Skin testing, including histamine and diluent controls, will be performed prior to and at one and four weeks after initiation of immunotherapy. At each time point, blood will be obtained to measure total and antigen-specific IgE levels, tryptase and cytokine levels, and basophil activation with the relevant allergens and C5a as a non-IgE-mediated control for basophil activation.

ELIGIBILITY:
Inclusion Criteria:

* Verified allergic sensitivity to either Timothy Grass or Short Ragweed pollen (primary allergen)
* Verified allergic sensitivity to at least one allergen in addition to the primary allergen

Exclusion Criteria:

* Negative skin testing to Timothy Grass or Short Ragweed pollen and at least one other environmental allergen
* Dermatographism
* Severe dermatologic condition that may interfere with skin testing
* Pregnancy
* H1 receptor antihistamine taken within 7 days of testing
* Systemic steroids
* Omalizumab taken at any time in the past
* Receiving or received allergen immunotherapy
* Desensitized to any drug within 6 months
* Current uncontrolled or severe asthma
* Eosinophilic esophagitis
* Significant pulmonary, cardiovascular, renal, hepatobiliary, or neurological diseases, or another disease process felt to put a subject at increased risk for adverse events
* Hypersensitivity to any of the inactive ingredients in the allergen extract tablets
* History of mental illness or drug or alcohol abuse that could interfere with the ability to comply with study requirements
* Inability or unwillingness to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-01-18 (Actual); Study Completion 2018-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence B Schwartz, M.D.,Ph.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhao W, Gomez G, Macey M, Kepley CL, Schwartz LB. In vitro desensitization of human skin mast cells. J Clin Immunol. 2012 Feb;32(1):150-60. doi: 10.1007/s10875-011-9605-8. Epub 2011 Oct 19. PMID 22009002
- [Background] Maloney J, Bernstein DI, Nelson H, Creticos P, Hebert J, Noonan M, Skoner D, Zhou Y, Kaur A, Nolte H. Efficacy and safety of grass sublingual immunotherapy tablet, MK-7243: a large randomized controlled trial. Ann Allergy Asthma Immunol. 2014 Feb;112(2):146-153.e2. doi: 10.1016/j.anai.2013.11.018. Epub 2013 Dec 21. PMID 24468255
- [Background] Creticos PS, Maloney J, Bernstein DI, Casale T, Kaur A, Fisher R, Liu N, Murphy K, Nekam K, Nolte H. Randomized controlled trial of a ragweed allergy immunotherapy tablet in North American and European adults. J Allergy Clin Immunol. 2013 May;131(5):1342-9.e6. doi: 10.1016/j.jaci.2013.03.019. PMID 23622121
- [Background] Cockcroft DW, Davis BE, Boulet LP, Deschesnes F, Gauvreau GM, O'Byrne PM, Watson RM. The links between allergen skin test sensitivity, airway responsiveness and airway response to allergen. Allergy. 2005 Jan;60(1):56-9. doi: 10.1111/j.1398-9995.2004.00612.x. PMID 15575931
- [Background] Niederberger V, Laffer S, Froschl R, Kraft D, Rumpold H, Kapiotis S, Valenta R, Spitzauer S. IgE antibodies to recombinant pollen allergens (Phl p 1, Phl p 2, Phl p 5, and Bet v 2) account for a high percentage of grass pollen-specific IgE. J Allergy Clin Immunol. 1998 Feb;101(2 Pt 1):258-64. doi: 10.1016/s0091-6749(98)70391-4. PMID 9500760

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After enrollment, allergen skin prick testing was performed to confirm sensitization to the required allergens. Of the 58 subjects enrolled, 37 were determined to lack sensitization to timothy grass pollen or ragweed pollen, plus at least one other environmental allergen. These subjects were excluded from the study prior to randomization. One subjected qualified, but was lost to follow up prior to randomizing.
Period: Overall Study
Arm/Group | Sublingual Allergen Tablets | Placebo
Started | 10 | 10
Completed | 10 | 9
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: One subject in placebo arm was lost to follow up and not analyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sublingual Allergen Tablets | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 2 | 2 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in PC3
Description: Change in the dose of allergen eliciting a wheal 3 mm greater than negative control upon skin prick testing (PC3)
Time Frame: Assessed at 2 weeks and at the end of the study (2 months)
Population: One subject from placebo arm not analyzed due to missing data
Measure: Median (Inter-Quartile Range); unit: Change in log dilution of allergen
Arm/Group | Sublingual Allergen Tablets | Placebo
Number analyzed (Participants) | 10 | 8
Change in log dilution of allergen | -0.2750 [-1.5900 to -0.0200] | -0.0250 [-0.5275 to 0.2500]

2. Primary Outcome: Change in Basophil Activation
Description: Change in the dose of allergen eliciting a 50% increase in number of basophils positive for CD63 and/or CD203c relative to negative and positive controls
Time Frame: Assessed at 2 weeks and at the end of the study (2 months)
Measure: Median (Inter-Quartile Range); unit: Change in log dilution of allergen
Arm/Group | Sublingual Allergen Tablets | Placebo
Number analyzed (Participants) | 10 | 9
Change in log dilution of allergen | -4.1100 [-7.8050 to -0.7050] | 0.1300 [-1.9275 to 2.9600]

3. Secondary Outcome: Cross-desensitization - PC3
Description: Change in the dose of an unrelated allergen eliciting a wheal 3 mm greater than negative control upon skin prick testing (PC3)
Time Frame: Assessed at 2 weeks and at the end of the study (2 months)
Measure: Median (Inter-Quartile Range); unit: Change in log dilution of allergen
Arm/Group | Sublingual Allergen Tablets | Placebo
Number analyzed (Participants) | 10 | 9
Change in log dilution of allergen | -0.0350 [-1.0250 to 0.3600] | 0.8000 [-0.1950 to 1.5175]

4. Secondary Outcome: Cross-desensitization - Basophil Activation
Description: as for outcome 2
Time Frame: Assessed at 2 weeks and at the end of the study (2 months)
Measure: Median (Inter-Quartile Range); unit: Change in log dilution of allergen
Arm/Group | Sublingual Allergen Tablets | Placebo
Number analyzed (Participants) | 10 | 9
Change in log dilution of allergen | -0.2000 [-2.3825 to 0.3075] | -0.1500 [-5.6625 to 0.7050]

5. Other Pre Specified Outcome: Percent Allergen-specific IgE
Description: The percent of total serum IgE that is specific for the primary allergen will be compared to the degree (if any) of cross-desensitization seen by skin prick or basophil activation testing
Time Frame: Assessed at enrollment, at 2 weeks, and at the end of the study (2 months)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for a total of 2 months while subjects were on treatment/placebo.
Arm/Group | Sublingual Allergen Tablets | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 1/10 | 0/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sublingual Allergen Tablets (N=10) | Placebo (N=9)
Throat irritation and ear fullness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-04-25): https://cdn.clinicaltrials.gov/large-docs/65/NCT02676765/Prot_SAP_000.pdf